CLINICAL TRIAL: NCT03399617
Title: Effect of an Innovative Behavioral Change Strategy and SQ-LNS on Stunting and Obesity in Children Living in Baja Verapaz, Guatemala
Brief Title: SPOON: Sustained Program for Improving Nutrition - Guatemala
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inter-American Development Bank (Other)
Collaborators: The PepsiCo Foundation (Other); Fundazúcar (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Inter-AmericanDB Guatemala
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Exclusive Breast Feeding; Feeding Patterns; Stunting; Obesity, Childhood
Keywords: Stunting; Obesity; Lipid-based Nutrient Supplements (LNS); Latin America; Child nutrition; Feeding practices
MeSH Terms: conditions — Breast Feeding; Feeding Behavior; Growth Disorders; Pediatric Obesity; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Care+MNPs (Active Comparator): Participants will receive standard health care services provided by the Ministry of Health, including micronutrient powders (MNPs). Children 6 months old will receive 1 gram of powdered micronutrients for 60 days every 6 months until 24 months of age.
  Interventions: Dietary Supplement: Micronutrient Powders
- SPOON behavioral change strategy+SQ-LNS (Experimental): Participants will receive Small Quantity Lipid-based Supplements (SQ-LNS) from 6-24 months and a behavioral change to promote adequate infant and young child feeding practices and the use of SQ-LNS will be delivered to mothers or caregivers. The behavioral change strategy includes individual home-visits, group sessions, and community mobilization activities. SQ-LNS consists of a 20g nutrient supplement package to be consumed daily from 6-24 of age. SQ-LNS formulation does not include sugar.
  Interventions: Behavioral: SPOON behavioral change strategy; Dietary Supplement: SQ-LNS
- SPOON behavioral change strategy+MNPs (Experimental): Participants will receive micronutrient powders (MNPs) from 6-24 months and a behavioral change to promote adequate infant and young child feeding practices and the use of MNPs will be delivered to mothers or caregivers. The behavioral change strategy includes individual home-visits, group sessions, and community mobilization activities.
  Interventions: Dietary Supplement: Micronutrient Powders; Behavioral: SPOON behavioral change strategy

INTERVENTIONS:
Dietary Supplement: Micronutrient Powders — Micronutrient powders (5 nutrient formulation) are currently provided by the Guatemalan Ministry of Health to children between 6-24 months of age.
  Other Names: MNPs
  Arms: SPOON behavioral change strategy+MNPs; Standard Care+MNPs
Behavioral: SPOON behavioral change strategy — An innovative behavioral change strategy designed using ethnographic and marketing methods to promote adequate infant and young child feeding practices and the use of SQ-LNS. The strategy will be delivered to mothers or caregivers through individual home-visits, group sessions, and community mobilization activities.
  Arms: SPOON behavioral change strategy+MNPs; SPOON behavioral change strategy+SQ-LNS
Dietary Supplement: SQ-LNS — SQ-LNS is a peanut-based ready to use home fortification product to improve diet quality in children 6-24 months of age. It includes peanuts and other ingredients such as vegetable fat, powdered milk and several micronutrients. The formulation designed for this study does not include sugar.
  Other Names: Smal Quantity Lipid-base Nutrient Supplements
  Arms: SPOON behavioral change strategy+SQ-LNS

SUMMARY:
The primary goal of this study is to assess the impact of an innovative strategy to prevent undernutrition and obesity in early childhood in children 0-24 months in Guatemala. This study is designed to evaluate the impact of promoting adequate infant an young child feeding practices and the use of SQ-LNS (Small Quantity Lipid-Based Nutrient Supplements) on the nutritional status of infants and young children. The study will be conducted in Baja Verapaz, Guatemala in conjunction with Fundazucar, Guatemala.

DETAILED DESCRIPTION:
SPOON Guatemala is an innovative strategy to prevent undernutrition and obesity in children aged 0-24 months living in high-poverty areas of Guatemala. SPOON focuses on improving feeding practices for infant and young children, including exclusive breastfeeding, and promote the use of home-fortification with peanut-based SQ-LNS (small quantity lipid-based nutrient supplements) through a novel behavior change strategy.

The study will recruit children between 0 and 3 months of age as well as pregnant women in the third trimester. Mothers or caregivers of eligible children will be invited to participate and a consent form obtain. Participation will start at 0-6 months and the intervention will last until children are 24 months. Participants will be randomly assigned at the community level to one of two groups: a control group and a treatment group. Participants in the control group will receive the standard services provided by their local health clinics in addition to a supply of micronutrient powders from 6-24 months of age, according to the national protocol. Participants in the treatment group will be randomly assigned at an individual level to receive two different interventions:

Treatment 1: This group will receive SQ-LNS supplement from 6-24 months and an innovative behavioral change strategy designed using ethnographic and marketing methods to promote adequate infant and young child feeding practices and the use of SQ-LNS. The strategy will be delivered to mothers or caregivers through individual home-visits, group sessions, and community mobilization activities.

Treatment 2. This group will receive micronutrient powders from 6-24 months and an innovative behavioral change strategy designed using ethnographic and marketing methods to promote adequate infant and young child feeding practices and the use of SQ-LNS. The strategy will be delivered to mothers or caregivers through individual home-visits, group sessions, and community mobilization activities.

A sample size of 500 children per group has been calculate to detect a minimum effect size of 0.2 with 95% level of significance and a 80% power for use of SQ-LNS. Additionally, a sample size of 40 communities and 500 children per group has been calculated to detect a minimum detectable effect size of 0.32 for communication.

Main outcomes include infant and young child feeding practices, height, weight, hemoglobin, prevalence of anemia, prevalence of stunting, prevalence of obesity, and weight gain rate. A baseline and final survey will be conducted to collect data for these variables, as well as sociodemographic information. Impact estimation will be done comparing the average results and the distribution of indicators between the treatment and control group. Differences of simple means and regression models including co-variables of the child's age and sex, and characteristics of the primary caregiver and household will be estimated. In addition to potential changes in indicator averages, changes in the distribution of variables will be explored under the hypothesis that the intervention might not only improve average value for a given indicator, but compress the distribution over a range of values closer to an optimal range. Changes to distributions will be checked by applying the Kolmogorov-Smirnov test.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in the third trimester or children 3 months of age
* Living in the defined intervention areas
* Children with no chronic diseases or congenital malformations
* Not planning on moving far from the intervention area in the next 24 months

Exclusion Criteria:

* Children with any chronic disease or congenital malformation
* Caretakers of the children plan on moving in the next 24 months
* Children with severe acute malnutrition

Max Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1280 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-12-18 (Actual)

PRIMARY OUTCOMES:
Infant and young child feeding practices | Measured at baseline and after 24 months of intervention
  Set of indicators of infant and young child feeding practices obtained by interview to participant mothers or caregivers
Height | Measured at 6 and 24 months of age
  Height-for-age z score obtained by measuring the height of participant children
Weight gain rate | Constructed from weight measurements at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, and 24 months of age
  Rate of weight gain from 0-24 months of age
Hemoglobin | Measured at 6 and 24 months of age
  Measurement of hemoglobin using a portable photometer
Prevalence of obesity in children | Measured at 6 and 24 months of age
  Population estimation of obesity using Population estimation of obesity using Body Mass Index (BMI)
Prevalence of stunting | Measured at 6 and 24 months of age
  Population estimation of stunting using height-for age <-2 SD
Prevalence of anemia | Measured at 6 and 24 months of age
  Population estimation of anemia using hemoglobin

SECONDARY OUTCOMES:
Adherence to Nutritional Supplement Regime | Measured every months from 6 months of age until the end of the intervention
  Consumption of the nutritional supplement measured as the number of packets consumed in one month
Exclusive Breastfeeding | Measured 24 months after the start of the intervention
  Measured as an indicator of exclusive breastfeeding, self-reported by the mother of a child

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Martinez, Study Director — IDB Evaluation Specialist
Locations (1):
- SPOON Guatemala, Rabinal, Departamento de Baja Verapaz, Guatemala

IPD SHARING:
Plan to Share IPD: Yes
Unidentified individual data will be shared among participating research institutions and made public 2 years after finalizing the study
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 2 years after finalizing the study
Access Criteria: Public

REFERENCES:
- [Derived] Gonzalez Acero C, Martinez S, Perez-Exposito A, Winters S. Effect of an innovative behavioural change strategy and small-quantity lipid-based nutrient supplements on stunting and obesity in children in Baja Verapaz, Guatemala: protocol for a randomised control trial. BMJ Open. 2020 Jul 19;10(7):e035528. doi: 10.1136/bmjopen-2019-035528. PMID 32690508